CLINICAL TRIAL: NCT04514601
Title: A Quality Improvement Project to Assess and Refine the Handover Process at Morning Trauma Meetings
Status: Completed | Type: Observational
Sponsor: Sandwell & West Birmingham Hospitals NHS Trust (Other)
Responsible Party: Principal Investigator, Salman Sadiq, Foundation Year 2 Doctor, Sandwell & West Birmingham Hospitals NHS Trust
Other Study IDs: QIP Trauma Meetings Sandwell
Record Dates: First submitted 2020-08-06; First posted 2020-08-17 (Actual); Last update posted 2020-08-17 (Actual); Status verified 2020-08

CONDITIONS: Neck of Femur Fracture; Fractures, Bone; Orthopedic Disorder
MeSH Terms: conditions — Femoral Neck Fractures; Fractures, Bone; Musculoskeletal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pre-Intervention Group: The verbal and written handover of these patients was observed. This included 146 general orthopaedic admissions patients and 43 trauma patients. All patient data was anonymised.
- Post-Intervention Group: The verbal and written handover of these patients was observed after the introduction of the intervention. This included 81 general orthopaedic admissions patients and 47 trauma patients. All patient data was anonymised.
  Interventions: Other: Standard Operating Protocol

INTERVENTIONS:
Other: Standard Operating Protocol — This was a written protocol on how the handover process should be conducted.
  Groups: Post-Intervention Group

SUMMARY:
This project was intended to observe the handover of trauma and orthopaedic patients at a district general hospital in the UK. Following the implementation of a standard operating protocol, the handover of patient information improved including neck of femur fracture patients significantly. The study can therefore be utilised by other similarly structured departments to improve the handover process, thereby improving patient safety.

DETAILED DESCRIPTION:
Poor handover and inadequate transmission of clinical information between shifts can result in patient harm. This study was designed to evaluate the impact of implementing a handover protocol on the quality of information exchanged in the trauma handover meetings in a UK hospital.

A prospective single centre observational study was performed at an acute NHS trust, using the Plan-Do-Study-Act (PDSA) methodology. Ten consecutive weekday trauma meetings, involving 43 patients, were observed to identify poor practices in handover. This data was used in conjunction with the Royal College of Surgeon's recommendations for effective handover (2007) to create a standard operating protocol (SOP). Following the implementation of the SOP, a further 8 consecutive weekday trauma meetings, involving a further 47 patients, were observed. The data collection was performed by 5 trained independent observers. The data was analysed using t test for quantitative variables and chi-square or Fisher's exact tests for categorical variables.

ELIGIBILITY:
Inclusion Criteria:

* All patients that were handed over were included in the study.

Exclusion Criteria:

* Nil.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Trauma and Orthopaedic patients.
Sampling Method: Probability Sample
Enrollment: 317 (Actual)
Dates: Start 2019-10-23 (Actual); Primary Completion 2019-12-13 (Actual); Study Completion 2019-12-13 (Actual)

PRIMARY OUTCOMES:
To assess the efficacy of the handover of trauma patients going to theatre. | Up to 6 weeks.
  A calculation was performed of how many patients had information handed over to the day staff. This included if a patient's past medical history, investigation results, plan, consent status, mark status and starvation status was handed over either written or verbally. This was expressed as a percentage.
To assess the handover of neck of femur (NOF) fracture patients. | Up to 6 weeks.
  A calculation was performed of how many patients with NOF fractures had information handed over. This included the patient's age, mechanism of injury, past medical history, investigation results, plan, consent status, mark status, starvation status, scoring system calculation and discussion with next of kin regarding resuscitation status. For each of these domains for each patient, if the information was handed over, this was noted and was expressed as a percentage.
To determine if unwell patients were being handed over from the admissions list or patients already on the ward. | Up to 6 weeks.
  From the handover meetings that were observed, it was noted whether 'unwell' patients from the ward had been handed over. This was expressed as a percentage from all the meetings that were observed.

CONTACTS AND LOCATIONS:
Overall Officials: Collette Samuels, Study Director — Audit Co-Ordinator Sandwell Hospital
Locations (1):
- Sandwell Hospital, West Bromwich, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided